CLINICAL TRIAL: NCT06767826
Title: The Effect of Care Based on the Salutogenesis Model on Coping With Stress and the Sense of Integrity in Preventing Digital Game Addiction in Adolescents
Brief Title: The Effect of Care Based on the Salutogenesis Model
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Eda Albayrak Günday, Research Assistant Doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ErciyesUnı1
Record Dates: First submitted 2024-07-18; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Supportive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): For the pre-test data, the Introductory Information Form, DOBÖ-7, EBÇÖ and BDİ were applied to the intervention group. After the pre-test, 45-60 minute sessions will be held once a week through home visits to the adolescents in the intervention group and an 8-week individual care program specific to each individual will be applied. In this program, the sense of integrity, digital game addiction and what addiction brings to life will be addressed in the first two weeks, the needs and requirements of the adolescents will be determined and care will be provided to the adolescents in line with the salutogenesis model and the care guide adapted to digital game addiction.
  Interventions: Behavioral: Salutogenesis Models
- Control (No Intervention): The adolescents in the control group will be introduced in the guidance room at school, explanations will be made and pre-test data will be taken. For the pre-test data, the Introductory Information Form, DOBÖ-7, EBÇÖ and BÖ will be applied to the control group. No intervention will be made to the adolescents in the control group throughout the process, their education at school will continue. If the adolescents have questions about the data forms, they will be answered. After the pre-test application, DOBÖ-7, EBÇÖ and BÖ will be applied to the adolescents again in the 3rd and 6th months. The 3rd month follow-up and 6th month follow-up measurements of the adolescents will be completed in the guidance room at school. The "handbook for preventing digital game addiction in adolescents" will be given to the control group at school after the 6th month follow-up measurement.

INTERVENTIONS:
Behavioral: Salutogenesis Models — On the basis of the Salutogenesis Model, this study is based on the development of individuals' internal and external resources for game addictions and strengthening their sense of integrity. It has been determined that digital game addiction and problematic internet use in adolescents form the basis of seven problems. These problems have been identified as mental health, vision, pain, sleep and rest patterns, nutrition, social contact and physical activity. Encouraging behavioral changes regarding internet use and teaching adolescents how to deal with these problems becomes a necessity in today's technology. In the literature, counseling has been provided for families and adolescents to prevent digital game addiction in adolescents.
  Arms: Experiment

SUMMARY:
On the basis of the Salutogenesis Model, this study is based on the development of individuals' internal and external resources for game addictions and strengthening their sense of integrity. It has been determined that digital game addiction and problematic internet use in adolescents form the basis of seven problems. These problems have been identified as mental health, vision, pain, sleep and rest patterns, nutrition, social contact and physical activity. Encouraging behavioral changes regarding internet use and teaching adolescents how to deal with these problems becomes a necessity in today's technology. In the literature, counseling has been provided for families and adolescents to prevent digital game addiction in adolescents. Care based on the salutogenesis model has never been studied in the world, but in Turkey, Uzdil et al. used the model in patient care by adapting it to care. Additionally, studies have suggested designing school-based intervention programs to prevent and reduce digital game addiction. In this context, the aim of the study is to improve coping with stress and eliminate digital game addiction by strengthening the sense of integrity of Care Based on the Salutogenesis Model in Preventing Digital Game Addiction in Adolescents.

DETAILED DESCRIPTION:
The internet, which is the most indispensable technology of today, appeals to the needs of all age groups, as well as highlighting individuality, being easily accessible almost always, giving a feeling of superiority and achievement, and being able to be played without being tied to a physical location. With its features, it constantly attracts the attention of adolescents and causes them to actively use the internet. Problems associated with high levels of gaming and internet use are increasingly recognized as a potential public health burden across the developed world. Digital game addiction is considered a mental health problem by the World Health Organization (2018) and the American Psychiatric Association, and the fact that adolescence is full of excitement, anxiety and stressors for adolescents makes them an important risk group in digital game addiction. It is seen in international studies that this risk among adolescent individuals is up to 17%. In the study conducted by Ay on 865 adolescents in our country, this rate was found to be 28.8%, which is a remarkable finding. Other studies support these rates and reveal that digital game addiction is high in adolescents. In addition, in a study conducted in our country during the pandemic period, when digital game playing times before the pandemic and during the pandemic were compared; It was determined that this period increased significantly during the pandemic process.

Since adolescence constitutes the bond between childhood and adulthood, the individual in this period where some changes occur in cognitive, physical, psychological and social terms brought about by the transition period; They face many stressors such as family relationships, friendship relationships, characteristics of the developmental period, society's expectations, and anxiety about passing the university exam. Adolescents; It has been reported that in order to cope with these stressors or escape from stress, there may be behavior of escaping from the real world and turning to the virtual world, and it may evolve into addiction as a result of increased gaming behavior due to a sustaining stress factor such as a negative parental attitude. Looking at international and national research, it is seen that adolescents with high stress levels have high levels of digital game addiction.

One of the models based on stress management is the Salutogenesis Model. Antonovsky introduced the sense of cohesion as a salutogenic concept to explain how and why people can cope with stress better. The model argues that the individual's ability to successfully manage many stressors is achieved through the development of a sense of integrity. Sense of integrity; It explains the individual's ability to cope with tension, use internal and external resources to solve his problems in a healthy way, and the individual's general stance towards problems. A low sense of integrity indicates that the person cannot cope with stressful situations and does not use appropriate coping strategies. In this context, it is noteworthy that there are no studies examining the sense of integrity of adolescents who are in a stressful developmental period and aiming to increase the sense of integrity.

The concept of a sense of wholeness as a result of the developmental process during adolescence indicates that the concept is viewed primarily as a result of individual life experiences, learning processes, and environmental influences, rather than as a primary source and determinant of positive health. As they grow and convey positive coping experiences, adolescents develop a general sense of intelligibility and manageability of demands and a sense of meaningfulness about life as it is and overcoming challenges. From this perspective, adolescence is seen as vital life stages that are crucial for the development of a sense of personal harmony and individual health biography.

On the basis of the Salutogenesis Model, this study is based on the development of individuals' internal and external resources for game addictions and strengthening their sense of integrity. It has been determined that digital game addiction and problematic internet use in adolescents form the basis of seven problems. These problems have been identified as mental health, vision, pain, sleep and rest patterns, nutrition, social contact and physical activity. Encouraging behavioral changes regarding internet use and teaching adolescents how to deal with these problems becomes a necessity in today's technology. In the literature, counseling has been provided for families and adolescents to prevent digital game addiction in adolescents. Care based on the salutogenesis model has never been studied in the world, but in Turkey, Uzdil et al. used the model in patient care by adapting it to care. Additionally, studies have suggested designing school-based intervention programs to prevent and reduce digital game addiction. In this context, the aim of the study is to improve coping with stress and eliminate digital game addiction by strengthening the sense of integrity of Care Based on the Salutogenesis Model in Preventing Digital Game Addiction in Adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Having education at high school level,
* Volunteer to participate in the study,
* Having received at least 13 to 35 points from the digital game addiction scale using the polythetic method,
* Having no history of psychiatric illness in his/her CV,
* Does not have aphasia or any other problem that may prevent communication, students will be included in the research.

Exclusion Criteria:

* Previously participated in a care program based on the salutogenesis model,
* Students with a digital game addiction scale score below 13 points will not be included in the study.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
stress coping skills in adolescents | 3 months after the pre-test application to the intervention group (in the 1st month after the maintenance program), 6-month follow-up purposes. The adolescents' 3rd month follow-up and 6th month
  The highest score that can be obtained in active and avoidant coping styles is 12 points and in negative coping style is 9 points, while the lowest score is 0 in all subscales. The higher the score of a coping strategy, the more actively it is used.

SECONDARY OUTCOMES:
a sense of integrity in adolescents | 3 months after the pre-test application to the intervention group (in the 1st month after the maintenance program), 6-month follow-up purposes. The adolescents' 3rd month follow-up and 6th month
  Understandability (Items 2, 6, 8, 9, 11), manageability (Items 3, 5, 10, 13), and meaningfulness (Items 1, 4, 7, 12). Items 1, 2, 3, 7, and 10 of these items should be reversed. The scale items are Likert-type, scored from 1 to 7. The scale allows for a total score as well as using subscale scores. The total BDI score varies between 13 and 91. High scores obtained from the scale indicate that the person has a high sense of coherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Eda Albayrak Günday, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No